CLINICAL TRIAL: NCT01895855
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Efficacy Trial of a Single Dose Live Oral Cholera Vaccine, PXVX0200 CVD 103-HgR, in Preventing Cholera Following Challenge With Vibrio Cholerae 10 Days or 3 Months After Vaccination
Brief Title: Safety and Efficacy Challenge Study of Live Oral Cholera Vaccine Candidate,PXVX0200, to Prevent Cholera
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PXVX-VC-200-003
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PXVX0200 (Experimental): Biological: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 5x10^8 CFU
  Interventions: Biological: PXVX0200
- Placebo (Placebo Comparator): Biological: Placebo physiological saline
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: PXVX0200 — Single dose; liquid suspension after reconstitution with buffer; 5x10^8
  Arms: PXVX0200
Biological: placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if PXVX0200 is safe and effective in preventing cholera infection

DETAILED DESCRIPTION:
A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Efficacy Trial of a Single Dose of Live Oral Cholera Vaccine Candidate, PXVX0200 CVD 103-HgR Strain, in Preventing Cholera following Challenge with Vibrio cholerae O1 El Tor Inaba 10 Days or 3 Months after Vaccination in volunteers aged 18-45 years

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women,
* age 18 to 45 years inclusive;
* normal medical history and physical examination; and
* no clinically significant abnormalities from:
* urine dipstick for glucose, protein, and blood
* complete blood count,
* serum hepatic transaminases,
* total bilirubin (direct if abnormal),
* creatinine,
* electrolytes,
* albumin, or
* electrocardiogram.
* Women must have a negative pregnancy test.

Exclusion Criteria:

* travel to a cholera endemic area in the previous 5 years;
* abnormal stool pattern or regular use of laxatives;
* history of eating disorders (such as bulimia), anal or rectal disorders, allergy to tetracycline and/or ciprofloxacin;
* history of cholera or enterotoxigenic E. coli challenge or infection;
* current or recent antibiotic use;
* pregnancy or nursing;
* positive serology for HIV, hepatitis B antigen, or hepatitis C;
* any immunosuppressive medical condition;
* history of hospitalization for psychiatric illness or use of specific psychiatric drugs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarty, MD, Study Director — Emergent BioSolutions
Locations (3):
- United States (3):
  - University of Maryland Baltimore, Baltimore, Maryland
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen WH, Cohen MB, Kirkpatrick BD, Brady RC, Galloway D, Gurwith M, Hall RH, Kessler RA, Lock M, Haney D, Lyon CE, Pasetti MF, Simon JK, Szabo F, Tennant S, Levine MM. Single-dose Live Oral Cholera Vaccine CVD 103-HgR Protects Against Human Experimental Infection With Vibrio cholerae O1 El Tor. Clin Infect Dis. 2016 Jun 1;62(11):1329-1335. doi: 10.1093/cid/ciw145. Epub 2016 Mar 21. PMID 27001804
- [Result] Haney DJ, Lock MD, Gurwith M, Simon JK, Ishioka G, Cohen MB, Kirkpatrick BD, Lyon CE, Chen WH, Sztein MB, Levine MM, Harris JB. Lipopolysaccharide-specific memory B cell responses to an attenuated live cholera vaccine are associated with protection against Vibrio cholerae infection. Vaccine. 2018 May 11;36(20):2768-2773. doi: 10.1016/j.vaccine.2018.04.011. Epub 2018 Apr 11. PMID 29655627
- [Result] Haney DJ, Lock MD, Simon JK, Harris J, Gurwith M. Antibody-Based Correlates of Protection Against Cholera Analysis of a Challenge Study in a Cholera-Naive Population. Clin Vaccine Immunol. 2017 May 31;24(8):e00098-17. doi: 10.1128/CVI.00098-17. Online ahead of print. PMID 28566334
- [Derived] Hossain M, Islam K, Kelly M, Mayo Smith LM, Charles RC, Weil AA, Bhuiyan TR, Kovac P, Xu P, Calderwood SB, Simon JK, Chen WH, Lock M, Lyon CE, Kirkpatrick BD, Cohen M, Levine MM, Gurwith M, Leung DT, Azman AS, Harris JB, Qadri F, Ryan ET. Immune responses to O-specific polysaccharide (OSP) in North American adults infected with Vibrio cholerae O1 Inaba. PLoS Negl Trop Dis. 2019 Nov 19;13(11):e0007874. doi: 10.1371/journal.pntd.0007874. eCollection 2019 Nov. PMID 31743334
- [Derived] Islam K, Hossain M, Kelly M, Mayo Smith LM, Charles RC, Bhuiyan TR, Kovac P, Xu P, LaRocque RC, Calderwood SB, Simon JK, Chen WH, Haney D, Lock M, Lyon CE, Kirkpatrick BD, Cohen M, Levine MM, Gurwith M, Harris JB, Qadri F, Ryan ET. Anti-O-specific polysaccharide (OSP) immune responses following vaccination with oral cholera vaccine CVD 103-HgR correlate with protection against cholera after infection with wild-type Vibrio cholerae O1 El Tor Inaba in North American volunteers. PLoS Negl Trop Dis. 2018 Apr 6;12(4):e0006376. doi: 10.1371/journal.pntd.0006376. eCollection 2018 Apr. PMID 29624592

RESULTS

PARTICIPANT FLOW:
Groups:
- PXVX0200: Biological: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 2x10^8 to 2x10^9 CFU in a liquid suspension
Period: Overall Study
Arm/Group | PXVX0200 | Placebo
Started | 95 | 102
Completed | 95 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PXVX0200 | Placebo | Total
Number analyzed (Participants) | 95 | 102 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 102 | 197
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.5 [18 to 45] | 30.6 [18 to 45] | 31.0 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 46 | 73
  Male | 68 | 56 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 89 | 97 | 186
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 64 | 69 | 133
  White | 26 | 32 | 58
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 95 | 102 | 197

OUTCOME MEASURES:

1. Primary Outcome: % of Participants With Moderate to Severe Diarrhea
Description: Determine whether a single dose of PXVX0200 provides significantly greater protection than placebo against a challenge with virulent V. cholerae O1 El Tor Inaba at 10 days after vaccination. The primary endpoint was the occurrence of moderate or severe (>/= 3 liters) diarrhea.
Time Frame: Ten days after vaccination
Measure: Number; unit: percentage of participants
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 35 | 66
percentage of participants | 5.7 | 59.1
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; 35 participants were challenged 10 days after receiving PXVX0200. 66 participants were challenged either 10 days or 90 days after receiving placebo; Test type: Superiority — The lower, two sided 95% confidence bound on protective efficacy must be >/= 30%; Vaccine Efficacy = 90.3, 95.1% CI 1-sided [lower limit 62.7] — Confidence intervals for the protective vaccine efficacy (PE) estimates were calculated using the method of Farrington and Manning (Farrington 1990)

2. Primary Outcome: % of Participants With Moderate to Severe Diarrhea
Description: Determine whether a single dose of PXVX0200 provides significant greater protection than placebo against a challenge with virulent V. cholerae O1 El Tor Inaba at 3 months after vaccination. The primary endpoint was the occurrence of moderate or severe (>/= 3 liters) of diarrhea.
Time Frame: Ninety days after vaccination
Measure: Number; unit: percentage of participants
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 33 | 66
percentage of participants | 12.1 | 59.1
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; 33 participants were challenged 90 days after receiving PXVX0200. 66 participants were challenged either 10 days or 90 days after receiving placebo; Test type: Superiority — The lower, two sided 95% confidence bound on protective efficacy must be >/= 30%; Vaccine Efficacy = 79.5, 95.1% CI 1-sided [lower limit 49.9] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Total Weight of Diarrheal Stools Following the 10 Day Cholera Challenge
Description: Total weight (converted to volume) per subject of diarrheal stools measured from subjects with diarrhea following the 10 day cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to Treat population comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Median (Full Range); unit: mL
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 35 | 66
mL | 309 [154 to 18164] | 4524 [140 to 24374]
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0073, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Weight of Diarrheal Stools Following the 90 Day Cholera Challenge
Description: Total weight (converted to volume) per subject of diarrheal stools measured from subjects with diarrhea following the 90 day cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to Treat population comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Median (Full Range); unit: mL
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 33 | 66
mL | 603 [22 to 9950] | 4524 [140 to 24374]
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; 33 participants were challenge 90 days after receiving PXVX0200. 66 participants were challenged either 10 days or 90 days after receiving placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: % of Participants With Diarrhea of Any Severity Following a 10 Day Cholera Challenge
Description: Incidence of mild or worse (any severity) diarrhea following the 10 day cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to treat population comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Number; unit: % of participants
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 35 | 66
% of participants | 14.3 | 92.4
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Vaccine Efficacy = 84.5, 95% CI 2-sided [67.0 to 100.0] — Confidence interval for the protective vaccine efficacy (PE) estimates were calculated using the method of Farrington and Manning (Farrington 1990)

6. Secondary Outcome: % of Participants With Diarrhea of Any Severity Following a 90 Day Challenge
Description: Incidence of mild or worse (any severity) diarrhea following the 90 day cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to treat population comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Number; unit: % of participants
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 33 | 66
% of participants | 45.5 | 92.4
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Vaccine Efficacy = 50.8, 95% CI 2-sided [33.6 to 66.8] — Confidence interval for protective vaccine efficacy (PE) estimates were calculated using the method of Farrington and Manning (Farrington 1990)

7. Secondary Outcome: % of Participants With Fever Following the 10 Day Cholera Challenge
Description: Incidence of mild or worse fever following the 10 day cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to treat population comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Number; unit: % of participants
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 35 | 66
% of participants | 2.9 | 27.3
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0025, Fisher Exact

8. Secondary Outcome: % of Participants With Fever Following the 90 Day Cholera Challenge
Description: Incidence of mild or worse fever following the 90 day cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to treat population comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Number; unit: % of participants
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 33 | 66
% of participants | 6.1 | 27.3
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0159, Fisher Exact

9. Secondary Outcome: Number of Days With Fecal Shedding Following 10 Day Challenge
Description: Number of days of fecal shedding of wild type V. cholerae following 10 Day Challenge.
Time Frame: Through 10 Days post challenge
Population: Intent to treat (ITT) population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 35 | 66
Days | 0.0 [0.0 to 2.0] | 3.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Days With Fecal Shedding Following 90 Day Challenge
Description: Number of days of fecal shedding of wild type V. cholerae following 90 Day Challenge
Time Frame: Through 10 days following challenge
Population: Intent to treat (ITT) population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 33 | 66
Days | 2.0 [1.0 to 3.0] | 3.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: PXVX0200 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: # of Days With Positive Stool Culture Following 10 Day Cholera Challenge
Description: Total number of days with a positive stool culture following the 10 Day Cholera challenge.
Time Frame: Through 10 Days following challenge
Population: Intent to treat (ITT) comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- PVXV0200: Biological: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 2x108 to 2x109 CFU in a liquid suspension
Arm/Group | PVXV0200 | Placebo
Number analyzed (Participants) | 35 | 66
Days | 0.9 (1.20) | 3.3 (1.01)
Statistical Analysis 1: Comparison: PVXV0200 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: # of Days With Positive Stool Culture Following 90 Day Cholera Challenge
Description: Total number of days with a positive stool culture following 90 Day Cholera Challenge
Time Frame: Through 10 Days following challenge
Population: Intent to treat (ITT) comprising all subjects who were randomized and received either PXVX0200 vaccine or placebo.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | PVXV0200 | Placebo
Number analyzed (Participants) | 33 | 66
Days | 2.1 (1.41) | 3.3 (1.01)
Statistical Analysis 1: Comparison: PVXV0200 vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: % of Participants With Reactogenicity, Diarrhea, Fever or Unsolicited Adverse Events Following Vaccination
Description: Incidence and severity of signs and symptoms of reactogenicity such as diarrhea, and fever following vaccination (through Day 8).
  Incidence and severity of unsolicited adverse events following vaccination (through Day 29).
Time Frame: Following vaccination (Days 1 - 8) and to Day 29
Measure: Number; unit: % of participants
Groups:
- PVXV0200: Biological: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 2x10^8 to 2x10^9 CFU in a liquid suspension
Arm/Group | PVXV0200 | Placebo
Number analyzed (Participants) | 95 | 102
% of participants
  % of Subjects with Reactogenicity | 49.5 | 50.0
  % of Subjects with Diarrhea Symptoms | 1.1 | 3.0
  % of Subjects with Fever Symptoms | 2.2 | 1.0
  % of Subjects with Unsolicited AEs | 17.9 | 16.7

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events were recorded for each vaccine or placebo recipient from the day of vaccination through 28 days after vaccination or 28 days after challenge, whichever was later. SAEs and medically attended AEs were recorded through the end of the follow-up period (Day 181).
Groups:
- PVXV0200: Biological: PXVX0200
  Single dose; liquid suspension after reconstitution with buffer; 5x10^8 CFU.
Arm/Group | PVXV0200 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/95 | 2/102
Other Adverse Events (participants affected / at risk) | 17/95 | 17/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PVXV0200 (N=95) | Placebo (N=102)
Hospitalization (Surgical and medical procedures) | 0 | 1 — Placebo recipient 01047 was hospitalized for orthopedic surgery considered unrelated to vaccination.
Hyperkalemia (Renal and urinary disorders) | 0 | 1 — Placebo recipient 03019 developed potentially life-threatening hyperkalemia 3 days post-challenge and was considered unrelated to vaccination.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PVXV0200 (N=95) | Placebo (N=102)
Eye pain (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 4
Feeling abnormal (General disorders) | 0 | 1
Feeling Hot (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 1
Upper Respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Sports injury (Injury, poisoning and procedural complications) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days